CLINICAL TRIAL: NCT04558814
Title: Evaluation of Serum Galectin-9 Level in Systemic Lupus Erythematosus Patients and it's Association With Disease Activity and Organ Damage
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, RHAbdelrahman, Resident doctor, Assiut University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Galectin-9 in SLE
Record Dates: First submitted 2020-09-16; First posted 2020-09-22 (Actual); Last update posted 2020-09-25 (Actual); Status verified 2020-09

CONDITIONS: Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Systemic lupus erythematosus patients (Other): Evaluation of serum galectin-9 level
  Interventions: Diagnostic Test: Serum galectin-9 level
- Control group (Other): Evaluation of serum galectin-9 level
  Interventions: Diagnostic Test: Serum galectin-9 level

INTERVENTIONS:
Diagnostic Test: Serum galectin-9 level — Determining level of galectin-9 in sera of patients of SLE with different disease activity and organ affection and Sera of control group

SUMMARY:
Study aims to evaluate serum galectin-9 in systemic lupus erythematosus patients and determine it's correlation with overall disease process

DETAILED DESCRIPTION:
Systemic lupus erythematosus (SLE) is an autoimmune disease characterized by producing large quantities of antibodies directed against self-antigens, particularly double stranded DNA (dsDNA) and small nuclear RNA-binding proteins such as Ro, La, Sm, and nRNP.

SLE-associated autoantibodies and high serum interferon alpha (IFN-α) are two important heritable phenotypes in SLE which are thought to play a role in disease pathogenesis . The most remarkable feature of the anti DNA response is its association with immunopathologic events especially glomerulonephritis . Immune complexes containing DNA can promote the expression of interferon alpha (IFN-alpha) by a specialized population of dendritic cells known as plasmacytoid dendritic cells .

Activation of the type I interferon (IFN) system is associated with disease pathogenesis in SLE, with affected patients typically demonstrating high concentrations of type I IFN proteins . Overexpression of type I IFN-induced genes that includes hundreds of gene transcripts; which is termed interferon signature (IFNGS), has been observed in 60-80% of adults and the majority of children with SLE .

Galectin-9 (Gal-9) is recognized as a novel, easy to measure biomarker for type1 IFN signatures and galectin-9 could aid in clinical decision making in SLE as a marker for disease activity and organ damage.

Galectin-9 is expressed by T cells, macro-phages, fibroblasts, and endothelial cells, its secreted form is barely detected under physiological conditions, it plays an recognizable role in the regulation of inflammation and immune responses by down-regulating pro-inflammatory T cells.

ELIGIBILITY:
Inclusion Criteria:

* clinically diagnosed systemic lupus erythematosus patients.

Exclusion Criteria:

* Individuals with other autoimmune diseases: 1)rheumatoid arthritis patients 2)dermatomyositis 3)scleroderma 4)mixed connective tissue disease

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-01 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Evaluate serum galectin-9 level in SLE patients and compare it with the serum galectin-9 level in healthy controls. | One year
  Compare level of galectin-9 in SLE patients with that of healthy controls

SECONDARY OUTCOMES:
compare galectin-9 in SLE patients with active and inactive renal disease. | One year
  Comparison of marker level between patients with active renal disease and patients without a tive renal disease

CONTACTS AND LOCATIONS:
Overall Officials: Mona Hussein, Doctor, Principal Investigator

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Muslimov IA, Iacoangeli A, Eom T, Ruiz A, Lee M, Stephenson S, Ginzler EM, Tiedge H. Neuronal BC RNA Transport Impairments Caused by Systemic Lupus Erythematosus Autoantibodies. J Neurosci. 2019 Sep 25;39(39):7759-7777. doi: 10.1523/JNEUROSCI.1657-18.2019. Epub 2019 Aug 12. PMID 31405929
- [Result] Catalina MD, Bachali P, Geraci NS, Grammer AC, Lipsky PE. Gene expression analysis delineates the potential roles of multiple interferons in systemic lupus erythematosus. Commun Biol. 2019 Apr 23;2:140. doi: 10.1038/s42003-019-0382-x. eCollection 2019. PMID 31044165
- [Result] Kudose S, Santoriello D, Bomback AS, Stokes MB, D'Agati VD, Markowitz GS. Sensitivity and Specificity of Pathologic Findings to Diagnose Lupus Nephritis. Clin J Am Soc Nephrol. 2019 Nov 7;14(11):1605-1615. doi: 10.2215/CJN.01570219. Epub 2019 Oct 25. PMID 31653670
- [Result] Ronnblom L, Leonard D. Interferon pathway in SLE: one key to unlocking the mystery of the disease. Lupus Sci Med. 2019 Aug 13;6(1):e000270. doi: 10.1136/lupus-2018-000270. eCollection 2019. PMID 31497305
- [Result] Matta B, Barnes BJ. Coordination between innate immune cells, type I IFNs and IRF5 drives SLE pathogenesis. Cytokine. 2020 Aug;132:154731. doi: 10.1016/j.cyto.2019.05.018. Epub 2019 May 23. PMID 31130331
- [Result] Brohawn PZ, Streicher K, Higgs BW, Morehouse C, Liu H, Illei G, Ranade K. Type I interferon gene signature test-low and -high patients with systemic lupus erythematosus have distinct gene expression signatures. Lupus. 2019 Nov;28(13):1524-1533. doi: 10.1177/0961203319885447. Epub 2019 Oct 29. PMID 31660791
- [Result] Matsuoka N, Fujita Y, Temmoku J, Furuya MY, Asano T, Sato S, Matsumoto H, Kobayashi H, Watanabe H, Suzuki E, Kozuru H, Yastuhashi H, Migita K. Galectin-9 as a biomarker for disease activity in systemic lupus erythematosus. PLoS One. 2020 Jan 27;15(1):e0227069. doi: 10.1371/journal.pone.0227069. eCollection 2020. PMID 31986153
- [Result] Chen HY, Wu YF, Chou FC, Wu YH, Yeh LT, Lin KI, Liu FT, Sytwu HK. Intracellular Galectin-9 Enhances Proximal TCR Signaling and Potentiates Autoimmune Diseases. J Immunol. 2020 Mar 1;204(5):1158-1172. doi: 10.4049/jimmunol.1901114. Epub 2020 Jan 22. PMID 31969388
- [Result] Vilar KM, Pereira MC, Tavares Dantas A, de Melo Rego MJB, Pitta IDR, Pinto Duarte ALB, da Rocha Pitta MG. Galectin-9 gene (LGALS9) polymorphisms are associated with rheumatoid arthritis in Brazilian patients. PLoS One. 2019 Oct 10;14(10):e0223191. doi: 10.1371/journal.pone.0223191. eCollection 2019. PMID 31600237
- [Result] Petri M, Orbai AM, Alarcon GS, Gordon C, Merrill JT, Fortin PR, Bruce IN, Isenberg D, Wallace DJ, Nived O, Sturfelt G, Ramsey-Goldman R, Bae SC, Hanly JG, Sanchez-Guerrero J, Clarke A, Aranow C, Manzi S, Urowitz M, Gladman D, Kalunian K, Costner M, Werth VP, Zoma A, Bernatsky S, Ruiz-Irastorza G, Khamashta MA, Jacobsen S, Buyon JP, Maddison P, Dooley MA, van Vollenhoven RF, Ginzler E, Stoll T, Peschken C, Jorizzo JL, Callen JP, Lim SS, Fessler BJ, Inanc M, Kamen DL, Rahman A, Steinsson K, Franks AG Jr, Sigler L, Hameed S, Fang H, Pham N, Brey R, Weisman MH, McGwin G Jr, Magder LS. Derivation and validation of the Systemic Lupus International Collaborating Clinics classification criteria for systemic lupus erythematosus. Arthritis Rheum. 2012 Aug;64(8):2677-86. doi: 10.1002/art.34473. PMID 22553077